CLINICAL TRIAL: NCT03176368
Title: Coconut Oil as a Novel Approach to Managing Radiation-Induced Xerostomia: An Interventional Study
Brief Title: Coconut Oil: Managing Radiation-Induced Xerostomia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20170139-01H
Record Dates: First submitted 2017-05-01; First posted 2017-06-05 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Xerostomia
Keywords: dry mouth; coconut oil; radiation
MeSH Terms: conditions — Xerostomia | interventions — Coconut Oil; Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coconut Oil (Experimental): Through a interventional/cohort design, we propose to study the experience of coconut oil over a three month period, allowing patients to use Biotene© oral lubricant (or another product of their choice) as an alternative to coconut oil if they so prefer.
  Interventions: Other: Coconut Oil

INTERVENTIONS:
Other: Coconut Oil — Coconut Oil
  Other Names: Natural Product

SUMMARY:
This study will seek to assess the experience of using of coconut oil as an approach to managing radiation-induced xerostomia in patients previously treated for cancer in the head and neck. There is a high prevalence of radiation-induced xerostomia in this patient population, and the condition has significant negative impact on patients' quality of life. There is currently no agreed-upon standard of care for the treatment of this condition. Anecdotal evidence from patients and both physicians and allied healthcare providers suggests improvement in this condition with the use of coconut oil, but this has not previously been formally studied. We therefore propose a case series study to formally assess the tolerability and efficacy of coconut oil as an approach to managing radiation-induced xerostomia.

DETAILED DESCRIPTION:
Xerostomia, or dry mouth, is a common complication in patients treated with radiotherapy for cancer of the head and neck, having been cited as occurring to some degree in 60- 100% of patients. Radiation, either alone or in addition to surgery, is a mainstay in the treatment of head and neck cancer. The incidence and degree of xerostomia as a side-effect is proportional to both the dosage of radiation used, and the amount of salivary gland tissue included in the radiation field. The downstream effects of xerostomia are wide-ranging, and can include difficulty chewing, swallowing, impaired phonation, altered taste sensation, dental carries, oropharyngeal candidiasis, systemic malnutrition and weight loss. Several studies have demonstrated a significant negative impact of xerostomia on patient quality of life. With cancer of the head and neck being the sixth most commonly diagnosed cancer worldwide, the burden of xerostomia on both the healthcare system and patient quality of life should not be underestimated.

There is no single effective treatment for radiation-induced xerostomia. Current treatments are non-specific, and directed at alleviating symptoms. These include lifestyle modifications (such as discontinuation of smoking, dairy, and other dietary products that thicken saliva), artificial saliva preparations, and parasympathetic agents such as pilocarpine which stimulate saliva production. Artificial saliva preparations such as Biotene© oral lubricant are commonly used today. However many of these treatments have limited efficacy, are costly, and the use of pilocarpine in particular is associated with significant side-effects. Other therapies which have been studied but not definitively proven effective include acupuncture and hyperbaric oxygen. Submandibular gland transfer, first described in 2000 and subsequently demonstrated in 2001, has also been shown to be effective in preventing xerostomia, however is a highly specialized procedure which prolongs the length of surgery, with benefit in only a limited patient population. Of these potential treatments, certainly Biotene© is the most common method of alleviating xerostomia. Preliminary evidence in the form of a phase II study has demonstrated the efficacy of Biotene© in alleviating symptoms of xerostomia in patients who have undergone radiation for head and neck cancer. The use of Biotene© is common practice at our tertiary care hospital, The Ottawa Hospital (TOH) although it is not agreed upon as THE standard of care.

Coconut oil, defined by Health Canada as a natural health / food product, has been anecdotally suggested to ameliorate the symptoms of xerostomia following radiation treatment for head and neck cancer. This anecdotal evidence has been derived from discussion with both patients and healthcare providers at The Ottawa Hospital. Both patients and allied health care providers involved in the care of patients following radiation treatment for head and neck cancer have attested to the beneficial effects of coconut oil. However, the effects of coconut oil in the management of radiation-induced xerostomia in patients previously treated for cancer of the head and neck have not been formally studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed treatment for head and neck cancer at least 18 months prior to entry to the study.
* Patient has experienced xerostomia following completion of radiation treatment.
* Patient has received external beam radiation at a dose of at least 50 Gy to the head and neck.
* Patients able to read / understand English.
* Patients who are competent/willing to consent to the study.
* Patients willing to comply with protocol and study schedule.

Exclusion Criteria:

* Patient currently undergoing treatment for head and neck cancer.
* Patient has previously used coconut oil for the treatment of xerostomia.
* Patient with allergy/sensitivity to coconut.
* Patient cannot read/ understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
Subjective benefit | 3 months
  Our primary outcome of interest will be descriptive in nature, namely whether patients find subjective benefit from the use of coconut oil, as evidenced by its continued use throughout the study period. This will be appraised qualitatively by analyzing diary entries.

SECONDARY OUTCOMES:
Quality of Life | 3 months
  Mean changes in Quality of Life Scores as measured by the Xerostomia-related quality of life scale (XeQOLS).
  - Subjective changes in speech quality, dysphagia, and sleep quality.
Change in Activities of Daily Living as assessed clinically at follow up appointment and as measured by the Xerostomia-related quality of life scale (XeQOLS). | 3 months
  Sleep Quality
Speech as assessed clinically at follow up appointment and as measured by the Xerostomia-related quality of life scale (XeQOLS). | 3 months
  Quality of speech
Dysphagia as assessed clinically at follow up appointment and by way of the XeQOLS. | 3 months
  Degree
Coconut Oil | 2 weeks or more
  Quantity and Frequency of Use as determined by diary entries.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Johnson-Obaseki, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No